CLINICAL TRIAL: NCT02958826
Title: Determining the Impact of External Sensory Stimuli on Patient Preferences During Outpatient Surgery
Brief Title: Impact of Sensory Stimuli on Patient Preferences During Outpatient Surgery
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Nicholas J Golda, Medical Director-University of Missouri Dermatology Clinics, University of Missouri-Columbia
Other Study IDs: 2005623
Record Dates: First submitted 2016-11-02; First posted 2016-11-08 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No Smoke Evacuation: No Smoke Evacuation Group, anonymous questionnaire administered
  Interventions: Other: Questionnaire
- Smoke Evacuation: Smoke Evacuation Group, anonymous questionnaire administered
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Anonymous questionnaire asking patients about their experiences with surgical lights, surgical smoke, and surgical sounds during their outpatient procedure.

SUMMARY:
The purpose of this study is to determine the effect surgical lights, surgical smoke, and surgical sounds have on patient satisfaction with their outpatient Mohs surgical procedure.

DETAILED DESCRIPTION:
The purpose of this study is to determine the impact of external sensory stimuli on patient preferences during outpatient Mohs surgery. Study participants will be asked to complete a questionnaire after their procedure sharing their experience with surgical lights, surgical smoke, and surgical noise. All responses are anonymous.

ELIGIBILITY:
Inclusion Criteria:

* All adult (> 18 years old) patients presenting for Mohs surgery and reconstruction for the treatment of nonmelanoma skin cancer on the head and neck

Exclusion Criteria:

* Subjects not meeting inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (> 18 years old) patients presenting for Mohs surgery and reconstruction for the treatment of nonmelanoma skin cancer on the head and neck.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Golda, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Smoke Evacuation Group: Treatment group with smoke evacuation used during the entire procedure (Mohs and reconstruction).
- Control Group: Control group with sham smoke evacuation.
Period: Overall Study
Arm/Group | Smoke Evacuation Group | Control Group
Started | 80 | 80
Completed | 80 | 80
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smoke Evacuation Group | Control Group | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Categorical [Count of Participants; unit: Participants] — Population: Two participants did not respond to this question
  Participants
    number analyzed (Participants) | 79 | 79 | 158
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 27 | 24 | 51
    >=65 years | 52 | 55 | 107
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 10 participants did not answer this question
  Participants
    number analyzed (Participants) | 78 | 72 | 150
    Female | 22 | 20 | 42
    Male | 56 | 52 | 108
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Effect of Surgical Lights on Patient Preference
Description: Prior to leaving the office, immediately after patient has completed Mohs surgical procedure, they will complete the questionnaire asking about their experience with surgical lights.
Time Frame: Questionnaire administered immediately after patient has completed Mohs surgical procedure. Questionnaire response data will be compiled and presented upon completion of the study in approximately one year.
Measure: Number; unit: percentage of participants
Arm/Group | No Smoke Evacuation | Smoke Evacuation
Number analyzed (Participants) | 80 | 80
percentage of participants
  Did not notice lights | 37.7 | 46.8
  Were not bothered by lights | 0.00 | 1.3
  Experience would not be improved if lights changed | 0.00 | 1.3

2. Primary Outcome: Effects of Surgical Smoke on Patient Preference
Description: Prior to leaving the office, immediately after patient has completed Mohs surgical procedure, they will complete the questionnaire asking about their experience with surgical smoke.
Time Frame: as for outcome 1
Population: Frequency of participants.
Measure: Number; unit: percentage of participants
Arm/Group | Smoke Evacuation Group | Control Group
Number analyzed (Participants) | 80 | 80
percentage of participants
  Did Not Notice Smoke Smell | 71.8 | 41.6
  Were Not Bothered by Smoke Smell | 93.6 | 75.0
  Would Not be More Satisfied with Smoke Evacuation | 89.6 | 77.3

3. Primary Outcome: Effect of Surgical Sounds on Patient Preference
Description: Prior to leaving the office, immediately after patient has completed Mohs surgical procedure, they will complete the questionnaire asking about their experience with surgical sounds.
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | No Smoke Evacuation | Smoke Evacuation
Number analyzed (Participants) | 80 | 80
percentage of participants
  Did not notice sounds | 51.9 | 50.0
  Were not bothered by sounds | 90.9 | 88.2
  Would not be more satisfied if sounds reduced | 93.2 | 84.2

ADVERSE EVENTS:
Time Frame: Adverse data were collected on the day of surgery for the time required to complete the procedure and questionnaire
Arm/Group | Smoke Evacuation Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT02958826/Prot_SAP_000.pdf